CLINICAL TRIAL: NCT06824506
Title: Evaluation of Early Postoperative Pulmonary Complications That Can be Detected by Ultrasonography in Patients Undergoing Laparoscopic Cholecystectomy With Low-flow Anesthesia
Brief Title: Ultrasound for Postop Lung Issues in Low-Flow Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Özgür Cirik, Assoc. Prof., Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: SanatoryumEAH-AK-01
Record Dates: First submitted 2025-02-06; First posted 2025-02-13 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Atelectasis, Postoperative; Cholecystitis; Gallstone; Pulmonary Atelectasis
Keywords: lung ultrasound; low flow anesthesia; laparoscopic cholecystectomy
MeSH Terms: conditions — Pulmonary Atelectasis; Cholecystitis; Gallstones

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low-Flow Anesthesia Group: As this study is observational in nature, no interventions will be performed by the research team. The study will involve a single group, within which the incidence and prevalence of the outcomes will be assessed.
  Interventions: Other: No-intervention

INTERVENTIONS:
Other: No-intervention — No interventions will be performed by the research team.

SUMMARY:
Detecting possible atelectasis and other respiratory problems that may develop immediately after extubation via lung ultrasonography can reduce pulmonary complications by performing necessary interventions such as oxygen support, respiratory exercises, mobilization, and non-invasive mechanical ventilation applications at an early stage. In addition, although low-flow anesthesia is frequently used in daily anesthesia practice, publications showing the effects of its use in laparoscopic cholecystectomy operations on pulmonary complications are limited. On this occasion, this study can be presented as a contribution to the literature.

DETAILED DESCRIPTION:
Postoperative atelectasis is a common complication that can develop in all patients receiving general anesthesia. The frequency of atelectasis increases due to increased intraabdominal pressure, especially in laparoscopic surgeries performed with pneumoperitoneum. For this reason, in order to prevent postoperative complications related to the lungs, it is extremely important to recognize atelectasis at an early stage, as well as to recognize the mechanisms that will cause atelectasis and avoid them.

Lung ultrasonography (Lung USG) draws attention for the rapid, cheap, safe and reliable detection of postoperative atelectasis. The fact that it can be applied at the bedside and can be easily repeated makes this method valuable. In the literature and in daily practice, it is seen that anesthesiologists commonly apply inhalation anesthesia with different fresh gas flow (FGF) rates during general anesthesia.

As defined by Baker and Simionescu, in low-flow anesthesia, FGF varies between 0.5 and 1 liter per minute. It has been shown that all types of flow are safe with modern anesthesia machines.

This study aims to demonstrate the effect of low-flow anesthesia (LFA) on pulmonary complications and, in particular, atelectasis that may develop after laparoscopic cholecystectomy operations, using a non-invasive, rapidly applicable, and proven method such as Lung USG.

ELIGIBILITY:
Inclusion Criteria:

* Patients with informed consent
* Patients scheduled for laparoscopic cholecystectomy
* Patients with a Body Mass Index between 18-35 kg/m²
* Patients in the American Society of Anesthesiologist (ASA) 1-2-3 category

Exclusion Criteria:

* Patients with emergency surgery planned
* Patients with ASA 4 and above
* Patients with lung disease
* Patients who have undergone thoracic surgery
* Pregnancy
* Patients with a preoperative Lung Ultrasound Score of 2 or 3 in any lung region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases that meet the inclusion and exclusion criteria will be included in the study. Patients will be taken to the operating room after being preoperatively evaluated in the observation room. The patient's anesthetic management will be provided by another anesthesiologist who is not participating in the study and is responsible for the patient. Intraoperative data will be obtained from the patient's anesthesia follow-up form and the records of the anesthesia machine. When the patients arrive in the recovery room, postoperative ultrasonographic measurements and other evaluations will be performed and noted. This group will include patients who received general anesthesia using low-flow techniques during the intraoperative period.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative atelectasis | 1 hour peroperatively
  Incidence of postoperative atelectasis determined by lung ultrasonography in patients undergoing laparoscopic cholecystectomy with low-flow anesthesia

SECONDARY OUTCOMES:
incidence of other postoperative pulmonary complications | 1 hour peroperatively
  Other postoperative pulmonary complications that may develop and be detected by ultrasonography such as pneumothorax, pleural effusion, pulmonary edema

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Özgür CIRIK, MD, Principal Investigator — Ankara Ataturk Sanatorium Training and Research Hospital
Locations (1):
- Ankara Ataturk Sanatorium Research and Training Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No